CLINICAL TRIAL: NCT05652335
Title: Phase 1, First-in-Human, Dose Escalation Study of JNJ-79635322, a Trispecific Antibody, in Participants With Relapsed or Refractory Multiple Myeloma or Previously Treated AL Amyloidosis
Brief Title: A Study of JNJ-79635322 in Participants With Relapsed or Refractory Multiple Myeloma or Previously Treated Amyloid Light-chain (AL) Amyloidosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109234; 79635322MMY1001 (Other: Janssen Research & Development, LLC); 2022-001465-12 (EudraCT Number); 2023-503679-12-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma; Previously Treated Amyloid Light-chain (AL) Amyloidosis
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive JNJ-79635322. The dose will be escalated sequentially until the recommended phase 2 dose (RP2D) regimen(s) have been identified.
  Interventions: Drug: JNJ-79635322
- Part 2: Dose Expansion (Experimental): Participants will receive JNJ-79635322 at the RP2D regimen(s) determined in Part 1.
  Interventions: Drug: JNJ-79635322

INTERVENTIONS:
Drug: JNJ-79635322 — JNJ-79635322 will be administered as SC injection.

SUMMARY:
The primary purpose of this study is to identify the recommended phase 2 dose (RP2D[s]) and schedule(s) to be safe for JNJ-79635322 in Part 1 (dose escalation), and to characterize the safety and tolerability of JNJ-79635322 at the RP2D(s) selected and in disease subgroups in Part 2 (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

For participants with relapsed or refractory multiple myeloma:

* Have a documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Part 1: Have relapsed or refractory disease, have been treated with a proteasome inhibitor, immunomodulatory drug (IMiD) agent, and an anti-CD38-based therapy for the treatment of multiple myeloma (MM),and should have been treated with at least 3 prior lines of therapy, or are refractory to proteosome inhibitor, IMiD agent, and an anti-CD38-based therapy regardless of prior lines of therapy, Part 2: Have relapsed or refractory disease, have been treated with a PI, IMiD and an anti-CD38 based therapy
* Must have an Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Have measurable disease at screening as defined by at least 1 of the following: a) Serum M-protein level greater than or equal to (>=) 0.5 grams per deciliter (g/dL); or b) Urine M-protein level >=200 milligrams (mg)/24 hours; or c) Light chain multiple myeloma: Serum immunoglobulin (Ig) free light chain (FLC) >=10 milligrams per deciliter (mg/dL) and abnormal serum Ig kappa lambda FLC ratio; d) For participants without measurable disease in the serum, urine, or involved FLC, presence of 1 or more focus of extramedullary disease (EMD) which meets the following criteria: extramedullary plasmacytoma not contiguous with a bone lesion, at least 1 lesion >=2 centimeter [cm] (at its greatest dimension) diameter on whole body Positron Emission Tomography and Computed Tomography (PET-CT) Scans (or whole body magnetic resonance imaging [MRI] approved by sponsor), and not previously radiated (Part 2C participants are not required to have measurable disease)

For participants with previously treated AL amyloidosis:

* Initial histopathological diagnosis of amyloidosis
* Participant who is not a candidate for available AL amyloidosis therapy with established clinical benefit and should have received at least 3 cycles of 1 prior line of therapy or a total of at least 2 cycles of 2 or more prior lines of therapy for AL amyloidosis
* Measurable disease at screening defined by at least 1 of the following: serum involved free light chain (iFLC) >=50 mg/L or difference between involved and uninvolved free light chains (dFLC) >=50 mg/L, or serum m-protein >= 0.5 g/dL
* One or more organs impacted by systemic AL amyloidosis
* Left ventricular ejection fraction (LVEF) >=45%

Exclusion Criteria:

For participants with relapsed or refractory multiple myeloma:

* Central Nervous System (CNS) involvement or clinical signs of meningeal involvement of multiple myeloma. If either is suspected, brain magnetic resonance imaging (MRI) and lumbar cytology are required
* Active plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or primary light chain amyloidosis
* Received a cumulative dose of corticosteroids equivalent to greater than (>) 140 mg of prednisone within the 14-day period before the start of study treatment administration
* Prior antitumor therapy as follows, in the specified time frame prior to the first dose of study treatment: (proteasome inhibitor [PI] therapy or radiotherapy within 14 days, immunomodulatory drug (IMiD) agent therapy within 7 days, gene-modified adoptive cell therapy within 90 days [not applicable for Part 2C participants], or CD3-redirecting therapy within 21 days[not applicable for Part 2B or 2C participants])
* Prior allogeneic transplant within 6 months before the start of study treatment administration or autologous transplant within 12 weeks before the start of study treatment administration
* Live, attenuated vaccine within 4 weeks before the first dose of study treatment
* Non-hematologic toxicity from prior anticancer therapy that has not resolved to baseline levels or to Grade less than or equal to (<=) 1 (except alopecia, tissue post-RT fibrosis [any grade] or peripheral neuropathy to Grade <=3)
* The following medical conditions: pulmonary compromise requiring supplemental oxygen use to maintain adequate oxygenation, human immunodeficiency (HIV) infection, active hepatitis B or C infection, stroke or seizure within 6 months prior to first dose of study treatment, autoimmune disease, serious active viral or bacterial infection, uncontrolled systemic fungal infection, cardiac conditions (myocardial infarction <=6 months prior to enrollment, New York Heart Association stage III or IV congestive heart failure, et cetera)
* Part 2C: have progressive disease or refractory disease per IMWG after CAR-T administration

For participants with previously treated AL amyloidosis:

* CNS involvement or clinical signs of meningeal involvement of AL amyloidosis. If either is suspected, whole brain MRI and lumbar cytology are required
* Any form of non-AL amyloidosis, including but not limited to transthyretin (ATTR) amyloidosis
* Active plasma cell leukemia, Waldenstrom's macroglobulinemia, or POEMS syndrome
* Pulmonary compromise requiring supplemental oxygen use
* Any serious medical conditions such as: active viral, bacterial, fungal infection; active autoimmune disease; HIV infection, active hepatitis B or C infection, stroke or seizure within 6 months prior to first dose of study treatment, significant cardiovascular conditions
* Previous or current diagnosis of symptomatic multiple myeloma
* Macroglossia that impairs swallowing difficulty
* Received a cumulative dose of corticosteroids equivalent to > 140 mg of prednisone within the 14-day period before the start of study treatment administration
* Prior antitumor therapy within 21 days prior to the first dose of study treatment (PI therapy or radiotherapy within 14 days, IMiD agent therapy within 7 days, gene-modified adoptive cell therapy within 90 days, or CD3-redirecting therapy within 21 days)
* Prior allogeneic transplant within 6 months before the start of study treatment administration or autologous transplant within 12 weeks before the start of study treatment administration
* Live, attenuated vaccine within 4 weeks before the first dose of study treatment
* Non-hematologic toxicity from prior anticancer therapy that has not resolved to baseline levels or to <=1 (except alopecia, tissue post-RT fibrosis [any grade] or peripheral neuropathy to Grade <=3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2027-04-19 (Estimated); Study Completion 2028-08-07 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose-limiting Toxicity (DLT) | Up to 2 years 5 months
  DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Parts 1 and 2: Number of Participants with Adverse Events (AEs) by Severity | Up to 2 years 5 months
  An adverse event is any untoward medical occurrence in a clinical study participant that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from grade 1 (mild) to grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event.
Part 2: Number of Participants with Abnormalities in Laboratory Values | Up to 2 Years 5 months
  Number of participants with abnormalities in laboratory values (hematology and chemistry) will be reported.

SECONDARY OUTCOMES:
Serum Concentration of JNJ-79635322 | Up to 2 Years 5 months
  Serum samples will be analyzed to determine concentrations of JNJ-79635322.
Number of Participants with Presence of Anti-Drug Antibodies to JNJ-79635322 | Up to 2 Years 5 months
  Number of participants with presence of anti-drug antibodies to JNJ-79635322 will be reported.
Preliminary Anticancer Activity of JNJ-79635322 as Defined by International Myeloma Working Group (IMWG) 2016 Response Criteria | Up to 2 Years 5 months
  Preliminary anticancer activity of JNJ-79635322 will be assessed according to the International Myeloma Working Group (IMWG) 2016 response criteria.
Time to Response (TTR) as Defined by IMWG 2016 Response Criteria | Up to 2 Years 5 months
  TTR is defined as the time between date of first dose of study drug and the first efficacy evaluation at which the participant has met all criteria for partial response (PR) or better as defined by IMWG 2016 response criteria.
Duration of Response (DOR) as Defined by IMWG 2016 Response Criteria | Up to 2 Years 5 months
  DOR is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of progressive disease (PD), per IMWG 2016 response criteria, or death due to any cause, whichever occurs first.
Part 2: Time to Response (TTR) as Defined by International Amyloidosis Consensus Criteria | Up to 2 Years 5 months
  TTR is defined as the time between date of first dose of study drug and the first efficacy evaluation at which the participant has met all criteria for PR or better as defined by International Amyloidosis Consensus Criteria.
Part 2: Duration of Response (DOR) as Defined by International Amyloidosis Consensus Criteria | Up to 2 Years 5 months
  DOR is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of progressive disease (PD), per International Amyloidosis Consensus Criteria or death due to any cause, whichever occurs first.
Part 2: Preliminary Anticancer Activity of JNJ-79635322 as Defined by International Amyloidosis Consensus Criteria | Up to 2 Years 5 months
  Preliminary anticancer activity of JNJ-79635322 will be assessed according to the International Amyloidosis Consensus Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (29):
- United States (9):
  - City of Hope, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - University of California San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania Division of Hematology Oncology Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Belgium (3):
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - CHU de Liege, Liège
- France (4):
  - CHU Nantes, Nantes
  - CHU Lyon Sud, Pierre-Bénite
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Institut Claudius Regaud, Toulouse
- Japan (3):
  - Japanese Red Cross Medical Center, Shibuya City
  - Osaka University Hospital, Suita-shi
  - The Cancer Institute Hospital of JFCR, Tokyo
- Netherlands (3):
  - VUMC Amsterdam, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - UMC Utrecht, Utrecht
- Spain (5):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
- United Kingdom (2):
  - University College Hospital, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Pillarisetti K, Yang D, Luistro L, Yao J, Smith M, Vulfson P, Testa J Jr, Ponticiello R, Brodeur SR, Heidrich B, Packman K, Singh S, Attar RM, Elsayed YA, Philippar U. Ramantamig (JNJ-79635322), a novel T-cell-engaging trispecific antibody targeting BCMA, GPRC5D, and CD3, in multiple myeloma models. Blood. 2025 Oct 16:blood.2025030027. doi: 10.1182/blood.2025030027. Online ahead of print. PMID 41100731